CLINICAL TRIAL: NCT05265637
Title: Algorithm for Vertical Placement of Implantable Collamer Lens
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: Valley Laser Eye Centre (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JB-21-001
Record Dates: First submitted 2022-02-11; First posted 2022-03-03 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Myopia
Keywords: implantable collamer lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Implantation of the Visian ICL: Visian implantable collamer lens (ICL)
  Interventions: Device: Visian

INTERVENTIONS:
Device: Visian — Visian implantable collamer lens (ICL)

SUMMARY:
The objective is to develop and evaluate an algorithm for implantable collamer lens (ICL) sizing that uses high frequency ultrasound biomicroscopy (UBM) for vertical placement.

DETAILED DESCRIPTION:
This study is a single-arm, clinical evaluation study of vault height and refraction, after successful ICL implantation. Subjects will be assessed pre-operatively, operatively, at 1 week postoperatively, and 1, 3, and 6 months post-operatively. Clinical evaluations will include measurement of monocular and binocular visual acuity, manifest refraction, and vault height.

ELIGIBILITY:
Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in each study eye.

Inclusion Criteria:

* Presenting for uncomplicated ICL implantation, either toric or non-toric lens, with vertical placement of the ICL
* Gender: Males and Females.
* Age: 23 or older.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error)
* Potential postoperative visual acuity of (20/25 Snellen) or better in the study eye

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or study eye, the subject should not be enrolled in the study.

* Irregular astigmatism (e.g. keratoconus)
* Unstable refractive error
* Low endothelial cell count
* Anterior chamber depth <2.8mm
* Any cataract in operative eye or nontraumatic cataract in the fellow eye
* Narrow anterior chamber angles (Grade 2 or less)
* Difficulties comprehending written or spoken language
* Patient with physical or intellectual disability (e.g. Down's Syndrome, Parkinson's Disease; unable to fixate)
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity.
* Participation in any investigational drug or device trial within the previous 30 days prior to the start date of this trial (or currently participating).

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 23 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with myopic or myopic astigmatism, and a motivation for spectacle independence.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Vault height | 6 months
  Vault height at 6-months postoperatively
Cycloplegic refraction | 3 months
  Percentage of eyes that are within postoperative MRSE ± 0.5D

SECONDARY OUTCOMES:
Monocular uncorrected distance visual acuity (Snellen) | 6 months
  Monocular uncorrected distance visual acuity (4m) at 6 months postoperatively using a Snellen Chart
Binocular uncorrected distance visual acuity (Snellen) | 6 months
  Binocular uncorrected distance visual acuity (4m) at 6 months postoperatively using a Snellen chart
Residual astigmatism | 6 months
  Residual astigmatism (as measured by manifest refraction at distance)

CONTACTS AND LOCATIONS:
Overall Officials: John Blaylock, MD, Principal Investigator — Valley Laser Eye Centre
Locations (1):
- Valley Laser Eye Centre, Abbotsford, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No